CLINICAL TRIAL: NCT03854968
Title: Quality Control Of Home Mechanical Ventilated Patient Mechanical Ventilators. A Multicenter Study
Brief Title: Quality Control of Home Mechanical Ventilators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Jose M. Montserrat, Principal Investigator, Hospital Clinic of Barcelona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VENTEST_2017
Record Dates: First submitted 2019-02-15; First posted 2019-02-26 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Mechanical Ventilation
Keywords: Mechanical ventilation; Performance
MeSH Terms: interventions — Quality Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quality control (Experimental): The participants home mechanical ventilator will be tested in order to performe a quality control
  Interventions: Other: Quality control

INTERVENTIONS:
Other: Quality control — The performance of the home mechanical ventilator of all patients in the study will be evaluated with a portable device

SUMMARY:
A multicentre quality control survey of home mechanical ventilation in patients. The prescribed ventilation settings, the settings of the ventilator control panel and the actual performance of the ventilator will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Home mechanically ventilated
* >18 years

Exclusion Criteria:

* Pacients with servoventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Pressure | 20 minutes
  ventilator pressures

CONTACTS AND LOCATIONS:
Overall Officials: Josep M Montserrat, Prof, Principal Investigator — Hospital Clinic
Locations (1):
- Hospital Clinic, Barcelona, Spain